CLINICAL TRIAL: NCT03287765
Title: Evaluating the Relationship Between Tau PET Imaging and CSF Biomarkers of AD in Humans
Brief Title: Evaluating the Relationship Between Tau PET Imaging and CSF Biomarkers of AD (Alzheimer Disease) in Humans
Acronym: ADRCproj1
Status: Completed | Type: Observational
Sponsor: Tammie L. S. Benzinger, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Tammie L. S. Benzinger, MD, PhD, Professor of Radiology & Neurological Surgery, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: IND123119,Protocol F
Record Dates: First submitted 2016-10-31; First posted 2017-09-19 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Alzheimer Disease
Keywords: Dementia; Tauopathies; cognitive impairment; CNS Diseases; neurodegenerative disease
MeSH Terms: conditions — Alzheimer Disease; Dementia; Tauopathies; Cognitive Dysfunction; Central Nervous System Diseases; Neurodegenerative Diseases | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Experimental 18F-AV-1451
  Interventions: Drug: 18F-AV-1451

INTERVENTIONS:
Drug: 18F-AV-1451 — Participants will receive a single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807. For those who cannot tolerate the full exam, participants will receive single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807.
  Other Names: Flortauapir

SUMMARY:
The purpose of this research study is to evaluate a new radioactive compound used in positron emission tomography (PET) scans in identifying tau tangles (a certain protein that might be associated with Alzheimer's disease) in the brain, and if the amount of tau tangles in the brain has a relationship to cerebrospinal fluid (CSF) biomarkers and cognitive status.

This study involves a PET scans using the radioactive compound, F 18 T807 for measurement of tau deposition. This radioactive compound is not approved by the United States Food and Drug Administration (FDA). An MRI will be conducted if one has not been completed completed within the past 12 months under a related research study. Participants will be asked about their medical history, family history, surgical history, and current medications. We will evaluate history of traumatic brain injury (TBI) using the Ohio State University Traumatic Brain Injury Identification (OSU TBI-ID) Method. This will take approximately 10 minutes. Participants will be asked to undergo a Mini Mental State Examination (MMSE), which will last approximately 5-10 minutes.

Additionally, participants may be invited to undergo optional brain PET imaging with 2-deoxy-2-[18F]fluoro-D-glucose fludeoxyglucose (18F-FDG), for measurement of the cerebral metabolic rate of glucose consumption. At the time of the initial T807-PET study, participants will be asked if they are willing to undergo repeat T807-PET imaging at least 2 years after the initial study. This follow up study is optional, and participation in the study and initial T807-PET imaging will not be contingent on agreeing to the 2-year follow up study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants, at least 65 years of age.
2. Participant is willing to undergo a lumbar puncture (LP) or has previously undergone LP. LP will be conducted under IRB ID 201109100 (PI: Anne Fagan).
3. Participant is able and willing to undergo positron emission tomography (PET) and magnetic resonance imaging (MRI) of the brain.
4. Pre-menopausal women must have a negative urine pregnancy test within 24 hours preceding T807 drug administration.

Exclusion Criteria:

1. Has any condition that, in the Investigator's opinion, could increase risk to the participant, limit the participant's ability to tolerate the experimental procedures, or interfere with the collection/analysis of the data (for example, participants with severe chronic back pain might not be able to lie still during the scanning procedures).
2. Is deemed likely unable to perform the imaging procedures for any reason.
3. Has a history of Torsades de Pointes or is taking medications known to prolong or may prolong QT interval (refer to study's list of restricted medications).
4. Has known hypersensitivity to T807 or any of its excipients.
5. Contraindications to PET, PET-CT or MR (e.g. electronic medical devices, inability to lie still for long periods) that make it unsafe for the individual to participate.
6. Severe claustrophobia.
7. Currently pregnant or breast-feeding. -

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Under this study protocol, collaborating physicians and the Knight Alzheimer's Disease Research Center (ADRC) Clinical Core will refer participants to the Knight ADRC Research Imaging (KARI) Program for MR and PET imaging to evaluate tau distribution in the brains of cognitively normal and cognitively impaired individuals.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Examine the association among T807-PET measures of PHF-tau. | 5 years
Characterize the amount and spatial distribution of T807-PET measures in healthy aging. preclinical AD, and early symptomatic AD. | 5 years
Characterize the amount and spatial distribution of T807-PET measures in preclinical AD. | 5 years
Characterize the amount and spatial distribution of T807-PET measures in early symptomatic AD. | 5 years
Examine the association among T807-PET measures of concentrations of CSF biomarkers. and cognitive performance. | 5 years
Examine the association among T807-PET measures of cognitive performance. | 5 years

SECONDARY OUTCOMES:
Evaluate the change in T807-PET measures over time in asymptomatic amyloid-positive individuals and its association with changes in concentrations of CSF biomarkers. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Benzinger, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The Investigators may share the participant's data with other researchers that may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at Washington University, at other research centers and institutions, or industry sponsors of research. The Investigators may also share the research data with large data repositories (a repository is a database of information) for broad sharing with the research community. If the individual research data is placed in one of these repositories only qualified researchers will be able to look at the information.